CLINICAL TRIAL: NCT03185455
Title: Remote Surveillance of Postpartum Hypertension
Acronym: TextBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 825390
Record Dates: First submitted 2017-06-06; First posted 2017-06-14 (Actual); Results first posted 2019-06-20 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Hypertension in Pregnancy
Keywords: Hypertension; Pregnancy; Text
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension

STUDY DESIGN:
Intervention Model Description: The study will be a randomized, two arm trial. Patient will be randomized to usual one time office visit based blood pressure check or to text-message based remote surveillance for two weeks. Randomization will be performed using a computer generated sequence using REDCAP. Demographic information will be collected from those who decline randomization or are ineligible in order to assess patient characteristics of those willing to be randomized and who meet eligibility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Those randomized to the standard protocol for blood pressure monitoring will be scheduled for an office based nursing blood pressure visits 4-6 days postpartum. Care at this visit is based on a physician derived algorithm.
- Remote (text based) surveillance (Experimental): Those randomized to remote surveillance will be provided with electronic blood pressure monitors prior to discharge and instructed on their use. Every day, for two weeks post-discharge, patients will receive a standard text message in the morning from a HIPAA compliant automated monitoring system reminding them to text their blood pressure. They will be asked to send in one blood pressure a day at minimum. They may be asked to send in more depending on the blood pressure result and clinical algorithm. This system will provide timely responses to patient texts and create a physician derived response to elevated blood pressures based on a programmed algorithm. Additionally, for blood pressures that reach a dangerous threshold, a clinical provider will be alerted per the algorithm and contact the patient for further evaluation.
  Interventions: Other: Remote (text based) surveillance

INTERVENTIONS:
Other: Remote (text based) surveillance — Women with hypertensive disorders of pregnancy with access to a cell phone with unlimited text message capabilities will be randomized to either office visit blood pressure checks after discharge or receive a blood pressure cuff and text in blood pressures for two weeks postpartum using a standardized, HIPAA compliant, physician derived automated platform.
  Arms: Remote (text based) surveillance

SUMMARY:
Women with hypertensive disorders of pregnancy need postpartum blood pressure (BP) surveillance to detect persistent hypertension. Various barriers result in only 30% attendance at postpartum BP visits. A more effective strategy is needed. Women with hypertension of pregnancy will be randomized to either text-based monitoring or office visits. Those randomized to the intervention will receive a BP cuff and text in their BP to an automated, clinician derived, HIPAA compliant text-based algorithm.

DETAILED DESCRIPTION:
Hypertension is a leading cause of maternal morbidity, mortality and obstetrical readmissions. Peak blood pressure usually occurs 3-6 days postpartum, and is typically unaccompanied by warning symptoms. Although there is a clear need for effective and reliable blood pressure surveillance after delivery, there are significant obstacles to in-person visits in the immediate postpartum period, including sleep deprivation, newborn care, and transportation needs. These barriers have proven real as we observed only 30-50% attendance to office blood pressure visits following delivery. This proposal will investigate whether text-based communication between patients and providers is an effective alternative method for monitoring postpartum hypertension in at risk women.

Women with hypertensive disorders of pregnancy with access to a cell phone with unlimited text message capabilities will be randomized to either office visit blood pressure checks after discharge or receive a blood pressure cuff and text in blood pressures for two weeks postpartum using a standardized, HIPAA compliant, physician derived automated platform.

ELIGIBILITY:
Inclusion Criteria:

* Women with chronic hypertension, gestational hypertension, or preeclampsia who deliver at the Hospital of the University of Pennsylvania will be eligible to participate. All patients must be > 18 years old, able to speak and read English, have a hypertension diagnosis, and have access to a cell phone with unlimited text message capabilities.

Exclusion Criteria:

* Women without access to a cell phone with unlimited text message capabilities will be excluded from the study in order to eliminate barriers to participate in remote surveillance. However, we will track the number of women not eligible for this reason in order to understand generalizability in an urban population.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hirshberg A, Downes K, Srinivas S. Comparing standard office-based follow-up with text-based remote monitoring in the management of postpartum hypertension: a randomised clinical trial. BMJ Qual Saf. 2018 Nov;27(11):871-877. doi: 10.1136/bmjqs-2018-007837. Epub 2018 Apr 27. PMID 29703800

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Women randomized to the standard protocol for blood pressure monitoring will be scheduled for an office based nursing blood pressure visits 4-6 days postpartum. The date and time of the office appointment is specified in the discharge document and reviewed with the patient prior to discharge. Care at this visit is based on a physician derived algorithm.
- Remote (Text Based) Surveillance: Women randomized to the text-based surveillance arm will be given an automatic Omron© blood pressure cuff and instructed on use by research team members prior to discharge. Patients will be enrolled into the texting program platform developed through Way to Health. A starting introductory text message is sent by the Way to Health platform to the phone number provided on day of discharge. Patients receive reminders to text message their blood pressures twice daily for two weeks postpartum, starting on the day after discharge. Immediate feedback is provided to the patient based on a preprogrammed automated algorithm. The primary investigator is alerted with pre-specified severe range blood pressure values (systolic blood pressure > 160 mmHg or diastolic > 100 mmHg) via text message or email and care is escalated as needed based on the same outpatient algorithm used in the office.
  Remote (text based) surveillance: Women with hypertensive disorders of pregnancy with access to
Period: Overall Study
Arm/Group | Standard of Care | Remote (Text Based) Surveillance
Started | 103 | 103
Completed | 103 | 103
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Remote (Text Based) Surveillance | Total
Number analyzed (Participants) | 103 | 103 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (5) | 28 (6) | 28 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 103 | 206
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 73 | 68 | 141
  White | 25 | 28 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 103 | 103 | 206
Medicaid Insurance [Count of Participants; unit: Participants] | 61 | 59 | 120
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 31 [25.1 to 38.3] | 30.1 [24.3 to 33.8] | 30.2 [24.6 to 35.8]
Nulliparous [Count of Participants; unit: Participants] | 52 | 61 | 113
Pregestational diabetes [Count of Participants; unit: Participants] | 3 | 5 | 8
Gestational diabetes [Count of Participants; unit: Participants] | 8 | 6 | 14
Chronic hypertension without antihypertensive medication [Count of Participants; unit: Participants] | 7 | 9 | 16
Chronic hypertension with antihypertensive medication [Count of Participants; unit: Participants] | 6 | 5 | 11
Renal disease [Count of Participants; unit: Participants] | 5 | 5 | 10
Gestational age at diagnosis [Median (Inter-Quartile Range); unit: weeks] | 38 [36 to 39] | 38 [36 to 39] | 38 [36 to 39]
Gestational age at delivery [Median (Inter-Quartile Range); unit: weeks] | 38 [37 to 39] | 38 [37 to 39] | 38 [37 to 39]
Gestational hypertension/preeclampsia without severe features [Count of Participants; unit: Participants] | 68 | 63 | 131
Preeclampsia with severe features [Count of Participants; unit: Participants] | 22 | 25 | 47
Hemolysis Elevated Liver Enzymes Low Platelet syndrome [Count of Participants; unit: Participants] | 3 | 0 | 3
Superimposed preeclampsia [Count of Participants; unit: Participants] | 10 | 14 | 24
Eclampsia [Count of Participants; unit: Participants] | 0 | 1 | 1
Induction of labor [Count of Participants; unit: Participants] | 58 | 54 | 112
Cesarean delivery in labor [Count of Participants; unit: Participants] | 18 | 23 | 41
Planned cesarean delivery [Count of Participants; unit: Participants] | 16 | 10 | 26
Magnesium sulfate use [Count of Participants; unit: Participants] | 32 | 35 | 67
Live birth [Count of Participants; unit: Participants] | 100 | 100 | 200
Discharged on oral antihypertensive medication [Count of Participants; unit: Participants] | 19 | 24 | 43
Postpartum discharge day [Median (Inter-Quartile Range); unit: day] | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3]
Breastfeeding [Count of Participants; unit: Participants] | 72 | 71 | 143

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whose Blood Pressure Was Assessed in the First Ten Days Following Discharge
Description: the percentage of patients in which a single blood pressure is obtained in the first 10 days following discharge. Within the texting group, the percentage of patients in whom blood pressures values are obtained at 72 hours and 7-10 days postpartum, in accordance with American College of Obstetricians and Gynecologists recommendations, will be assessed as well.
Time Frame: 10 days postdischarge
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Remote (Text Based) Surveillance
Number analyzed (Participants) | 103 | 103
Participants | 45 | 95

2. Secondary Outcome: Number of Participants Who Required Antihypertensive Medication Initiation or Dose Adjustment Within 2 Weeks Postpartum
Description: Number of participants who required antihypertensive medication initiation or dose adjustment within 2 weeks postpartum
Time Frame: 2 weeks postpartum
Population: Only women who attended the office visit were analyzed in the standard of care group
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Remote (Text Based) Surveillance
Number analyzed (Participants) | 45 | 103
Participants | 10 | 17

3. Secondary Outcome: Number of Participants Who Required Additional ER or Office Visits for Hypertension (Not Resulting in Readmission) Within 2 Weeks Postpartum
Description: Number of participants who required additional ER or office visits for hypertension (not resulting in readmission) within 2 weeks postpartum
Time Frame: 2 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Remote (Text Based) Surveillance
Number analyzed (Participants) | 103 | 103
Participants | 2 | 3

4. Secondary Outcome: Number of Participants With Hypertension Related Readmission Within 2 Weeks Postpartum
Description: Number of participants with hypertension related readmission within 2 weeks postpartum
Time Frame: 2 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Remote (Text Based) Surveillance
Number analyzed (Participants) | 103 | 103
Participants | 4 | 0

5. Secondary Outcome: Patient Satisfaction
Description: Patient who would recommend the program to a family or friend as per the Patient Satisfaction Survey completed at 2 weeks postpartum.
Time Frame: 2 weeks postpartum
Population: The data population analyzed in the Remote Surveillance Arm included only those who completed the satisfaction survey. Participants in the standard of care arm were not eligible to complete the Patient Satisfaction Survey since they did not receive the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Remote (Text Based) Surveillance
Number analyzed (Participants) | 0 | 77
Participants | 0 | 77

ADVERSE EVENTS:
Time Frame: 6 weeks postpartum
Arm/Group | Standard of Care | Remote (Text Based) Surveillance
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/103
Other Adverse Events (participants affected / at risk) | 0/103 | 0/103

LIMITATIONS AND CAVEATS:
one model of obstetrical care blood pressure monitors were not wireless

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT03185455/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT03185455/ICF_001.pdf